CLINICAL TRIAL: NCT01649765
Title: A Multi-center, Randomized, Placebo-Controlled Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of Belimumab, a Human Monoclonal Anti-BLyS Antibody, Plus Standard Therapy in Pediatric Patients With Systemic Lupus Erythematosus
Brief Title: Pediatric Lupus Trial of Belimumab Plus Background Standard Therapy
Acronym: PLUTO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Human Genome Sciences Inc., a GSK Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114055; 2011-000368-88 (EudraCT Number)
Expanded Access: NCT03125486 (No longer available)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE Flare Index; SRI; belimumab; efficacy; safety; B lymphocyte; BLyS; SELENA SLEDAI; BILAG; Lupus; Systemic Lupus Erythematosus (SLE); PGA; Pharmacokinetics; placebo; PRINTO
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): belimumab 10mg/kg IV monthly
  Interventions: Drug: belimumab 10mg/kg
- Arm 2 (Placebo Comparator): Normal Saline IV monthly
  Interventions: Other: placebo

INTERVENTIONS:
Drug: belimumab 10mg/kg — belimumab 10mg/kg IV monthly
  Arms: Arm 1
Other: placebo — Normal Saline 250 ml
  Other Names: Normal Saline
  Arms: Arm 2

SUMMARY:
This is a multi-center study to evaluate the safety, pharmacokinetics, and efficacy of belimumab intravenous (IV) in pediatric patients 5 to 17 years of age with active systemic lupus erythematosus

DETAILED DESCRIPTION:
This is a multi-center study to evaluate the safety, pharmacokinetics, and efficacy of belimumab intravenous (IV) in pediatric patients 5 to 17 years of age with active systemic lupus erythematosus (SELENA SLEDAI score ≥ 6). The study will consist of three phases: a 52-week randomized, placebo-controlled, double-blind phase; a long term open label continuation phase; and a long term safety follow up phase. The long term open label continuation and safety follow up periods will continue for at least 5 years and possibly up to 10 years from a subject's initial treatment with belimumab. Enrolment will be staggered by age cohorts to allow safety and PK interim analyses. Subjects will be randomized to belimumab 10mg/kg or placebo IV monthly dosing while continuing to receive background standard therapy throughout the study. An independent data monitoring committee (IDMC) will monitor the study as it progresses.

ELIGIBILITY:
Inclusion Criteria:

* 5 years to 17 years of age at enrollment
* Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) classification criteria.
* Have active SLE disease (SELENA SLEDAI score ≥ 6).
* Have positive anti-nuclear antibody (ANA) test results.
* Are on a stable SLE treatment regimen at a fixed dose for a period of at least 30 days prior to Day 0.
* Females of childbearing age are willing to use appropriate contraception
* Subject age appropriate assent and parent or legal guardian informed consent to participate

Exclusion Criteria:

* Pregnant or nursing.
* Have received treatment with belimumab (BENLYSTA®) at any time. (BENLYSTA® is a registered trademark of the GSK group of companies.)
* Treatment with any B cell targeted therapy (for example, rituximab) or an investigational biological agent in the past year.
* Have received anti-TNF therapy; Interleukin-1 receptor antagonist; IVIG; or plasmapheresis within 90 days of Day 0.
* Have received high dose prednisone or equivalent (>1.5mg/kg/day) within 60 days of baseline.
* Have received intravenous (IV) cyclophosphamide within 60 days of Day 0.
* Have received any new immunosuppressive/immunomodulatory agent, anti-malarial agent within 60 days of baseline.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have had a major organ transplant.
* Have significant unstable or uncontrolled acute or chronic diseases or conditions not due to SLE.
* Have a planned surgical procedure.
* History of malignant neoplasm within the last 5 years.
* Have required management of acute or chronic infections in the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test, or test positive at screening for HIV, Hepatitis B, or Hepatitis C.
* Have an IgA deficiency.
* Have severe laboratory abnormalities.
* Have had anaphylactic reaction to X-ray contrast agents or biologic agents.
* Suicidal behavior or ideation.
* Children in Care(CiC): a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2028-04-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (7):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cincinnati, Ohio
- Argentina (3):
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Santa Fe
- Canada (2):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
- Japan (4):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, San Luis Potosí City, Mexico
- GSK Investigational Site, Lima, Peru
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Warsaw
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tolyatti
- Spain (3):
  - GSK Investigational Site, Esplugues de Llobregat. Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- United Kingdom (3):
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunner HI, Abud-Mendoza C, Viola DO, Calvo Penades I, Levy D, Anton J, Calderon JE, Chasnyk VG, Ferrandiz MA, Keltsev V, Paz Gastanaga ME, Shishov M, Boteanu AL, Henrickson M, Bass D, Clark K, Hammer A, Ji BN, Nino A, Roth DA, Struemper H, Wang ML, Martini A, Lovell D, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Safety and efficacy of intravenous belimumab in children with systemic lupus erythematosus: results from a randomised, placebo-controlled trial. Ann Rheum Dis. 2020 Oct;79(10):1340-1348. doi: 10.1136/annrheumdis-2020-217101. Epub 2020 Jul 22. PMID 32699034
- [Background] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Background] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 93 pediatric participants with Systemic Lupus Erythematosus (SLE) were enrolled at 29 study centers in 10 different countries. This was a multi-center study to evaluate the safety, efficacy and pharmacokinetics of belimumab plus background standard therapy. The results presented are based on Part A (double blind).
Pre-assignment Details: The study consisted of three separate phases: Randomized, placebo-controlled, double-blind 52-week treatment phase (Part A), Long term belimumab open label safety follow up for participants who completed Part A (Part B) and Long term safety follow-up phase for participants who were withdrawn from Part A or Part B at any time (Part C).
Groups:
- Placebo: Participants received saline infusion (placebo) intravenously monthly for 48 weeks on a background of standard of care.
- Belimumab 10 mg/kg: Participants received 10 milligrams per kilograms (mg/kg) reconstituted solution intravenously monthly for 48 weeks on a background of standard of care.
Period: Overall Study
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 40 | 53
Completed | 31 | 45
Not Completed | 9 | 8
Not completed — Adverse Event | 5 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 40 | 53 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (2.17) | 13.5 (2.59) | 14.0 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 49 | 88
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: White - White/Caucasian/European Heritage | 21 | 27 | 48
  Race customized: Asian | 6 | 8 | 14
  Race customized: African American/African Heritage | 2 | 3 | 5
  Race customized: American Indian or Alaskan Native | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With SLE Responder Index (SRI) Response at Week 52
Description: SRI response is defined as >=4 point reduction, from Baseline in safety of estrogen in lupus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) score, no worsening (increase of <0.30 points from Baseline) in physician's global assessment (PGA) and no new British Isles Lupus Assessment Group of SLE clinics (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with Baseline. Analysis was performed using a logistic regression model for the comparison between belimumab and placebo with covariates treatment group, Baseline SELENA SLEDAI score (<=12 vs. >=13). Percentage of participants with SRI response at Week 52 of Part A were reported. Intent-to-Treat Population comprised of all participants who were randomized and treated with at least one dose of study agent in Part A. One participant had missing data at Baseline and therefore, could not be included in the analysis.
Time Frame: Week 52
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 39 | 53
Percentage of participants | 43.6 | 52.8
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.64 to 3.46]

2. Secondary Outcome: Percentage of Participants Meeting Pediatric Rheumatology International Trials Organization (PRINTO)/ American College of Rheumatology (ACR) Juvenile SLE Response Evaluation Criteria for Improvement in Juvenile SLE at Week 52 Using Definition 1 and 2
Description: Percentage of participants meeting PRINTO/ACR Juvenile SLE Response Evaluation criteria for improvement in juvenile SLE using two different PRINTO/ACR Juvenile SLE Response Evaluation definitions of improvement that is Definition 1: At least 50% improvement in any 2 of 5 endpoints below and no more than 1 of the remaining worsening by more than 30% and Definition 2: At least 30% improvement in 3 of 5 endpoints below and no more than 1 of the remaining worsening more than 30%. Endpoints were: 1. Percent change in Parent's Global Assessment (ParentGA) at Week 52, 2. Percent change in PGA at Week 52, 3. Percent change in SELENA SLEDAI score at Week 52, 4. Percent change in Pediatric Quality of Life Inventory (PedsQL) physical functioning domain at Week 52, 5. Percent change in 24 hour proteinuria at Week 52 (gram/24hour equivalent by spot urine protein to creatinine ratio).
Time Frame: Week 52
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 40 | 53
Percentage of participants
  Definition 1 | 35.0 | 60.4
  Definition 2 | 27.5 | 52.8
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.15 to 6.54] — Definition 1
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority; Odds Ratio (OR) = 2.92, 95% CI 2-sided [1.19 to 7.17] — Definition 2

3. Secondary Outcome: Percent Change From Baseline in ParentGA at Week 52
Description: ParentGA assesses the participant's overall well-being at the moment rated on a 21-numbered circle visual analog scale (VAS; 0 - very well, 10 - very poorly). Baseline was defined as measurements at Day 0. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline value X 100. Last Observation Carried Forward (LOCF) was used. Eight participants had a score of zero at Baseline and therefore, could not be included in the analysis.
Time Frame: Baseline (Day 0) and Week 52
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 38 | 47
Percent change | -23.61 [-95.0 to 600.0] | -53.85 [-100.0 to 900.0]

4. Secondary Outcome: Percent Change From Baseline in PGA at Week 52
Description: The PGA is a 10 centimeter (cm) visual analogue scale (VAS), anchored at 0 (none) and 3 (severe), designed for the physician to indicate the participant's overall disease activity at a particular visit as part of the validated SELENA SLEDAI index. Primary investigator or a subinvestigator scored the PGA for the participant, and same person evaluated the participant each time. Baseline was defined as measurements at Day 0. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline value X 100. LOCF was used.
Time Frame: Baseline (Day 0) and Week 52
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 40 | 53
Percent change | -48.802 (42.0423) | -56.525 (43.7939)

5. Secondary Outcome: Percent Change From Baseline in SELENA SLEDAI at Week 52
Description: The SELENA SLEDAI score is a weighted index for assessing SLE disease activity in which signs and symptoms, laboratory tests and physician's assessment for each of 9 organ system were given a weighted score and summed if present at the time of the visit or in the preceding 10 days. A SELENA SLEDAI score of 0 would suggest no lupus activity; while a score of 105 is the maximum calculable if all items were scored as being present from active lupus. A decrease of 4 points or more equates to a clinically meaningful improvement. Baseline was defined as measurements at Day 0. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline value X 100. One participant had missing data at Baseline and therefore, could not be included in the analysis.
Time Frame: Baseline (Day 0) and Week 52
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 39 | 53
Percent change | -38.0 (39.50) | -43.3 (43.73)

6. Secondary Outcome: Percent Change From Baseline in PedsQL Physical Functioning Domain Score at Week 52
Description: The PedsQL is a generic quality of life scale validated for the pediatric population which consists of 23 items, encompassing 4 health domains: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items). From the raw scores of the 23 items, a total summary score and individual domain scores can be calculated. The total and domain scores are each transformed on a 0 to 100 score with higher scores indicating higher quality of life. For Physical Functioning Domain scale, score was from 0 to 100 where, 0 indicates lower quality of life and 100 indicates greater quality of life. Baseline was defined as measurements at Day 0. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline Value X 100. LOCF was used.
Time Frame: Baseline (Day 0) and Week 52
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 40 | 53
Percent change | 12.5 [-53 to 575] | 10.5 [-100 to 280]

7. Secondary Outcome: Percent Change From Baseline in Proteinuria at Week 52
Description: Percent change from Baseline in proteinuria was calculated. The percent change from baseline to Week 52 in 24 hour proteinuria was analyzed using summary statistics and 95% confidence intervals, without any adjustment for covariates. Baseline was defined as measurements at Day 0. Percent change from Baseline was calculated by subtracting the Baseline value from value at Week 52 divided by the Baseline Value X 100. LOCF was used.
Time Frame: Baseline (Day 0) and Week 52
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 40 | 53
Percent Change | 7.0920 [-90.568 to 570.149] | -2.1277 [-85.073 to 1681.884]

8. Secondary Outcome: Percentage of Participants With a Sustained SRI Response
Description: Sustained SRI response was defined as having a response on the primary efficacy endpoint at Weeks 44, 48, and 52. Data for percentage of participants with a sustained SRI response was presented. Drop Outs and Treatment Failures were considered Non-Responders. Only those participants with data available at specific time point were analyzed.
Time Frame: Up to 52 weeks
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 39 | 53
Percentage of participants | 41.0 | 43.4

9. Secondary Outcome: Percentage of Participants With a Sustained ParentGA Response
Description: Sustained ParentGA response was defined as having >0.7 improvement at Weeks 44, 48, and 52 compared at Baseline. Data for percentage of participants with a sustained ParentGA response was presented. Thirteen participants had a score of <=0.7 at Baseline and therefore, could not be included in the analysis.
Time Frame: Up to 52 weeks
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 36 | 44
Percentage of Participants | 33.3 | 59.1

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with AEs and SAEs have been reported.
Time Frame: Up to 60 weeks
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 40 | 53
Participants
  AEs | 33 | 42
  SAEs | 14 | 9

11. Secondary Outcome: Maximum Concentration at Steady State (Cmax, ss) and Minimum Concentration at Steady State (Cmin, ss)
Description: The pharmacokinetic (PK) population comprised all participants included in the As- Treated population for whom at least one post belimumab treatment PK sample was obtained and analyzed. The PK model was fitted to the observed serum concentration-time data. The maximum (Cmax) and minimum (Cmin) concentrations reported in this table are model derived values at ss, assuming a 10 mg/kg dose administered once every 28 days.
Time Frame: 28-days dosing interval at steady state
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 53
Micrograms per milliliter
  Cmax, ss | 315 (31.2)
  Cmin, ss | 50 (68.3)

12. Secondary Outcome: Area Under Curve of Belimumab at Steady State (AUC, ss)
Description: The PK model was fitted to the observed serum concentration-time data. The AUC values reported in this table are model derived values at ss, assuming a 10 mg/kg dose administered once every 28 days.
Time Frame: 28-days dosing interval at steady state
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 53
Micrograms per milliliter | 3012 (43.2)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from start of the study to the follow up visit (Up to 60 weeks).
Description: Intent-to-Treat Population was used to collect adverse events.
Arm/Group | Placebo | Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/53
Serious Adverse Events (participants affected / at risk) | 14/40 | 9/53
Other Adverse Events (participants affected / at risk) | 27/40 | 36/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Belimumab 10 mg/kg (N=53)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 2 (2)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Retinal vasculitis (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Belimumab 10 mg/kg (N=53)
Nasopharyngitis (Infections and infestations) | 8 (11) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 6 (8)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (6)
Pharyngitis (Infections and infestations) | 3 (3) | 3 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (3)
Urinary tract infection (Infections and infestations) | 4 (8) | 1 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (4) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 7 (9)
Nausea (Gastrointestinal disorders) | 3 (4) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 10 (17) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (10) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 4 (5) | 4 (4)
Pyrexia (General disorders) | 3 (10) | 2 (2)
Fatigue (General disorders) | 2 (4) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 3 (3)
Blood immunoglobulin G decreased (Investigations) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (3) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT01649765/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT01649765/SAP_001.pdf